CLINICAL TRIAL: NCT06630026
Title: Examining the Validity and Reliability of the Dresden Falls Questionnaire in Patients With Parkinson's Diagnosis Living in Turkey
Acronym: DREFAQ
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, PhD Research Assistant, Istanbul Medeniyet University
Other Study IDs: 2024/115 DREFAQ
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Falls; Scale Reliability Validity
Keywords: Parkinson disease; Falls; Scale reliability validity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson Patients: Parkinson patients who are aged 18-80 years with Hoehn & Yahr scale between 1-4 and able to speak and read Turkish, will recruit to the study.
  Interventions: Other: The aim of this study is to adapt the Dresden Falls Questionnaire scale (DREFAQ)scale to Turkish society in Parkinson patients and to make its validity and reliability in Turkish.

INTERVENTIONS:
Other: The aim of this study is to adapt the Dresden Falls Questionnaire scale (DREFAQ)scale to Turkish society in Parkinson patients and to make its validity and reliability in Turkish. — • The aim of this study is to adapt the Dresden Falls Questionnaire scale (DREFAQ)scale to Turkish society and to make its validity and reliability in Turkish. It has 5 questions. This study will be conducted with Parkinson patients. The patients will be sought to answer questionnaires during regular rehabilitation sessions.

SUMMARY:
The aim of this study is to adapt the Dresden Falls Questionnaire scale (DREFAQ) to Turkish society and to make its validity and reliability in Turkish. The DREFAQ) scale developed by Frank, Anika, et al assesses falls in patients with Parkinson. It has 5 questions. This study will be conducted with Parkinson patients. The patients will be sought to answer questionnaires during regular rehabilitation sessions. 50 participants will be included in the study. In order to evaluate the validity of the DREFAQ, the Modified Falls Efficacy Scale (MFES), which can evaluate the efficacy of falls and has been validated in Turkish, and the Parkinson's Disease Quality of Life (PDQOL) questionnaire, which can evaluate the quality of life and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

DETAILED DESCRIPTION:
The reliability and validity of the scale will begin with language equivalence and cultural adaptation. The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained from these two Turkish translations with a common opinion.

The scale, which has been translated into Turkish, will be translated into English by two other people who are fluent in Turkish and English. The scale translated into English will be compared with the original. If the developer of the scale, Frank, Anika, et al approves the translation of the scale, participants will be recruited for the study. In the pre-trial phase, a reassessment will be conducted with 15 participants to test the intelligibility of the scale. Based on the results of the pre-test phase, the final version of DREFAQ will be able to be modified. The data of DREFAQ are collecting through face-to-face when the patients came to the rehabilitation center. 50 participants will be included in the study.

In order to evaluate the validity of the DREFAQ, the Modified Falls Efficacy Scale (MFES), which can evaluate the efficacy of falls and has been validated in Turkish, and the Parkinson's Disease Quality of Life (PDQOL) questionnaire, which can evaluate the quality of life and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a Hoehn & Yahr score between 1-4,
* Individuals who can ambulate with or without assistive equipment,
* Individuals with a Mini Mental State Examination score of >24,
* Individuals with a history of falling at least once in the last year,

Exclusion Criteria:

* communication or cognitive problems,
* aphasia and speech disorders
* unstable medical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson patients who are aged 18-80 years with Hoehn & Yahr score between 1-4 and able to speak and read Turkish.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Falls | Baseline
  Falls will be assessed with the Dresden Falls Questionnaire scale (DREFAQ). DREFAQ consists of 5 items in total. Items 1 to 4 are scored from 0 to 3. The total score of the DREFAQ is calculated by summing the first 4 items (0-12). The location of the injury (from item 4) and the circumstances (item 5) are not used in the score calculation but provide additional qualitative information. Higher scores indicate a high risk of falling.
Falls Efficacy | Baseline
  Falls efficacy will be assessed with the Modified Falls Efficacy Scale (MFES) scale. The MFES consists of 14 items in total. Items are scored from 0 (not sure of himself/herself) to 10 (totally confident). Total score is between 0-140. Lower scores indicate a high risk of falling.

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQoL) | Baseline
  Ouality of life will be assessed with the Parkinson's Disease Quality of Life (PDQOL) questionnaire. It consists of 8 questions in total. Items are scored 0 to 4. Total score is between 0-32. Higher scores indicate lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No